CLINICAL TRIAL: NCT07372144
Title: Phase III, Randomized, Double-blind, Placebo-controlled Study Investigating the Efficacy of Creatine Supplementation in Attenuating Chemotherapy-related Cognitive Decline in Patients With Early-stage Breast Cancer Undergoing Chemotherapy.
Brief Title: Creatine and Cognitive Health in Patients With Early-stage Breast Cancer During and After Chemotherapy Treatment
Acronym: IARA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: D'Or Institute for Research and Education (Other)
Responsible Party: Principal Investigator, Renata Rodrigues da Cunha Colombo Bonadio, Doctor, Principal Investigator, D'Or Institute for Research and Education
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IARA NUP 25000.193607/2025-11
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study. Participants, investigators, study staff involved in clinical care, outcome assessment, cognitive testing, imaging analyses, laboratory analyses, and data analysis are masked to treatment allocation. Creatine and placebo are identical in appearance, taste, and packaging. Unblinding will occur only if required for participant safety, according to predefined protocol procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Placebo (Placebo Comparator): Participants assigned to this arm will receive a placebo powder matched in appearance, taste, and packaging to the investigational product. The placebo will be administered orally once daily, dissolved in water, starting 7 days before the first cycle of chemotherapy and continuing until 12 months after completion of chemotherapy.
  Interventions: Other: Placebo
- Arm B: Creatine Supplementation (Active Comparator): Participants assigned to this arm will receive oral creatine monohydrate at a dose of 5 g per day, dissolved in water and administered once daily. Treatment will begin 7 days before the first cycle of chemotherapy and will continue until 12 months after completion of chemotherapy.
  Interventions: Drug: Creatine

INTERVENTIONS:
Drug: Creatine — Oral creatine monohydrate supplementation administered at a fixed dose of 5 g per day, dissolved in water and taken once daily. The intervention starts 7 days before initiation of neoadjuvant or adjuvant chemotherapy and continues through chemotherapy and up to 12 months after chemotherapy completion. The intervention is designed to evaluate the preventive effect of creatine on chemotherapy-related cognitive impairment, with longitudinal cognitive, clinical, imaging, and translational assessments. The comparator is a matched placebo identical in appearance, taste, and packaging.
  Arms: Arm B: Creatine Supplementation
Other: Placebo — Oral placebo powder matched in appearance, taste, and packaging to the investigational product, administered once daily dissolved in water. The placebo is initiated 7 days before the start of neoadjuvant or adjuvant chemotherapy and continued through chemotherapy and up to 12 months after chemotherapy completion. The placebo contains no active ingredients and is used as the comparator to assess the preventive effect of creatine supplementation on chemotherapy-related cognitive impairment.
  Arms: Arm A: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate whether oral creatine supplementation can prevent chemotherapy-related cognitive impairment in patients with early-stage breast cancer undergoing neoadjuvant or adjuvant chemotherapy. The main questions it aims to answer are:

* Does creatine supplementation reduce the occurrence and severity of chemotherapy-related cognitive impairment, as measured by patient-reported cognitive function?
* Does creatine supplementation preserve objective cognitive performance compared with placebo during and after chemotherapy?

Researchers will compare creatine supplementation (5 g/day) with placebo to assess differences in cognitive outcomes, safety, and exploratory biological markers.

Participants will:

* Receive oral creatine or placebo starting 7 days before chemotherapy and continuing until 12 months after chemotherapy completion
* Complete patient-reported cognitive assessments and objective neuropsychological tests at predefined time points
* Undergo clinical follow-up for safety and oncologic outcomes
* Provide blood samples for biomarker analyses and stool samples for gut microbiota assessment
* Undergo brain magnetic resonance imaging at selected study visits

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Histologically confirmed invasive breast cancer (stages I-III).
* Indication for neoadjuvant or adjuvant chemotherapy containing an anthracycline or a taxane.
* Targeted therapies and hormone therapy are permitted according to clinical indication.
* Ability to provide informed consent and comply with study procedures.
* ECOG performance status 0-2.
* Ability to maintain adequate hydration.

Exclusion Criteria:

* Prior neurologic conditions that may impair cognitive assessment, including previous stroke, dementia, traumatic brain injury with neurologic sequelae, or other neurologic disorders affecting cognition.
* Uncorrected sensory impairments that preclude cognitive assessment and/or completion of study instruments.
* History of uncontrolled psychiatric disorders that may interfere with cognitive evaluation.
* Creatinine clearance <60 mL/min, calculated using the Cockcroft-Gault formula.
* Known liver disease.
* Pregnancy.
* Heart failure.
* Presence of ascites.
* Inflammatory bowel disease.
* Chronic use of nonsteroidal anti-inflammatory drugs (NSAIDs).
* Lactation.
* Chronic use of immunosuppressive agents, including doses greater than 10 mg/day or equivalent.
* Prior chronic creatine supplementation within the last 3 months.
* Known allergy to any component of the supplement or placebo.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in patient-reported cognitive function | Baseline and 1 month after completion of chemotherapy
  Measured by the Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog), version 3, from baseline to 1 month after completion of chemotherapy. A clinically significant cognitive decline is defined as a decrease of at least 7.5 points in the total FACT-Cog score.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto D'Or de Pesquisa e Ensino de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No